CLINICAL TRIAL: NCT02721979
Title: A Phase 2 Study of Apalutamide in Active Surveillance Patients
Brief Title: Apalutamide in Treating Patients With Prostate Cancer Who Are in Active Surveillance
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual
Sponsor: University of Washington (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Schweizer, Assistant Professor, Division of Medical Oncology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9582; NCI-2016-00221 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9582 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1716037 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2016-03-11; First posted 2016-03-29 (Estimated); Results first posted 2021-03-29 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (apalutamide) (Experimental): Patients receive apalutamide PO QD for 90 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Apalutamide; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; JNJ 56021927; JNJ-56021927
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well apalutamide works in treating patients with prostate cancer who are in active surveillance. Testosterone can cause the growth of prostate cancer cells. Hormone therapy using androgen receptor antagonist apalutamide may fight prostate cancer by blocking the use of testosterone by the tumor cells.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive apalutamide orally (PO) once daily (QD) for 90 days in the absence of disease progression or unacceptable toxicity.

After completion of the study treatment, patients are followed up at 180, 365, 545, and 730 days; and at years 3, 4 and 5 by medical record review.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an informed consent document
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
* Written authorization for use and release of health and research study information has been obtained
* Life expectancy >= 10 years (as determined by the treating physician)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Histologically confirmed adenocarcinoma of the prostate as documented by a minimum 12 core prostate biopsy completed within 1-year of enrollment (note: most recent prostate biopsy must have demonstrated prostatic adenocarcinoma)
* Favorable risk prostate cancer as defined by:

  * Very low-risk:

    * Clinical stage T1c disease
    * PSA density (PSAD) < 0.15 ng/mL
    * Gleason score 6
    * =< 2 core biopsies with =< 50% involvement of any biopsy core with cancer, or unilateral disease =< 2 core biopsies with any percentage involvement OR
  * Low risk:

    * Clinical stage =< T2a
    * PSA < 15 ng/mL
    * Gleason score 6 OR
  * Low-intermediate risk:

    * Clinical stage T1c
    * PSA < 15 ng/ml
    * Gleason 3+4 present in =< 50% of one core/site as detected by systematic biopsy or MRI/transrectal ultrasound (TRUS) fusion guided biopsy
    * Gleason 6 disease in all other cores / sites
* Willing and qualified for active surveillance at Johns Hopkins or the University of Washington
* Serum testosterone >= 150 ng/dL
* Able to swallow the study drugs whole as a tablet
* Hemoglobin >= 9.0 g/dL, (at screening), independent of transfusion and/or growth factors within 3 months prior to registration
* Platelet count >= 100,000 x 10^9/uL (at screening) independent of transfusion and/or growth factors within 3 months prior to registration
* Serum albumin >= 3.0 g/dL (at screening)
* Glomerular filtration rate (GFR) >= 45 mL/min (at screening)
* Serum potassium >= 3.5 mmol/L (at screening)
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN) (at screening) (note: in subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject may be eligible)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 × ULN (at screening)
* Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to study entry
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug; must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Prior local therapy to treat prostate cancer (e.g. radical prostatectomy, radiation therapy, brachytherapy)
* Prior use of ARN-509 (apalutamide)
* Have known allergies, hypersensitivity, or intolerance to ARN-509 (apalutamide) or its excipients
* Prior or ongoing systemic therapy for prostate cancer including, but not limited to:

  * Hormonal therapy (e.g. leuprolide, goserelin, triptorelin)
  * Cytochrome P450 (CYP)-17 inhibitors (e.g. abiraterone, ketoconazole)
  * Antiandrogens (e.g. bicalutamide, nilutamide)
  * Second generation antiandrogens (e.g. enzalutamide)
  * Immunotherapy (e.g. sipuleucel-T, ipilimumab)
  * Chemotherapy (e.g. docetaxel, cabazitaxel)
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements
* History of any of the following:

  * Seizure or known condition that may pre-dispose to seizure (including but not limited to prior stroke, transient ischemic attack, loss of consciousness within 1 year prior to registration, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
  * Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to registration
  * Any condition that in the opinion of the investigator, would preclude participation in this study
* Current evidence of any of the following:

  * Uncontrolled hypertension
  * Gastrointestinal disorder affecting absorption
  * Active infection (e.g. human immunodeficiency virus [HIV] or viral hepatitis) or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
  * Any condition that in the opinion of the investigator, would preclude participation in this study
* The use of drugs known to lower the seizure threshold, including: atypical antipsychotics (e.g. clozapine, olanzapine, risperidone, ziprasidone), bupropion, lithium, meperidine, pethidine, phenothiazine antipsychotics (e.g. chlorpromazine, mesoridazine, thioridazine), and tricyclic antidepressants (e.g. amitriptyline, desipramine, doxepin, imipramine, maprotiline, mirtazapine)
* The use of strong CYP3A4 inhibitors, including: itraconazole, clarithromycin, erythromycin, diltiazem, verapamil, delavirdine, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, grapefruit juice (or grapefruits)

  * Note: If a patient is on a strong CYP3A4 inhibitor, they can be reconsidered for enrollment if they can safely stop said medication; a two week or 5 half-lives, whichever is longer, washout will be required prior to enrolling on study; subject may not resume medication while receiving apalutamide
* Strong CYP3A4 inducers, including: phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, efavirenz, tipranavir, St. John's wort

  **Note: If a patient is on a strong CYP3A4 inhibitor, they can be reconsidered for enrollment if they can safely stop said medication; a two week or 5 half-lives, whichever is longer, washout will be required prior to enrolling on study; subject may not resume medication while receiving apalutamide
* Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schweizer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The screening study procedures are conducted within 30 days prior to enrollment. The only exception to this would be the surveillance prostate biopsy.
Pre-assignment Details: 24 subjects signed consent for this study, but only 23 were eligible to enter into the treatment phase.
Groups:
- Apalutamide: Day 1 until Day 90. Patients receive apalutamide PO QD for 90 days in the absence of disease progression or unacceptable toxicity.
  Apalutamide: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Apalutamide
Started | 23
Completed | 22
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: There are 24 participants who signed the consent form, and only 23 progressed into the treatment phase. One patient was a screen fail.
Arm/Group | Treatment (Apalutamide)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24
Patients with very low risk disease at baseline [Count of Participants; unit: Participants] — Patients deemed to have very low risk disease based on NCCN criteria at the time of enrollment. Population: Only patients that did not screen fail are included in this analysis.
  Participants
    number analyzed (Participants) | 23
    (all) | 9

OUTCOME MEASURES:

1. Primary Outcome: Negative (i.e. no Residual Carcinoma) Site Directed and Systematic Prostate Biopsy Rate
Description: Negative rate will be presented as the percent of subjects with a negative repeat biopsy, and will be calculated as: (number of patients with a negative biopsy following 90-days of apalutamide) / (total number of patients enrolled on the study) x 100. A 1-sample chi-square test will be used to compare the proportion with a negative repeat biopsy to the null hypothesis value of 20% (above). The 95% confidence interval will be computed.
Time Frame: At 90 days
Population: These are patients that had 90 days of treatment and had post-treatment biopsies.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Apalutamide
Number analyzed (Participants) | 22
percentage of subjects | 59 [37 to 78]

2. Secondary Outcome: Percentage of Patients Exiting Active Surveillance Due to Pathologic Reclassification
Description: The percentage of patients who exited active surveillance due to pathologic reclassification (e.g. increasing tumor volume or gleason score) will be computed along with its 95% confidence interval.
Time Frame: At 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment (Apalutamide)
Number analyzed (Participants) | 22
Percentage of participants | 18.2 [6.6 to 41.2]

3. Secondary Outcome: Percentage of Patients Exiting Active Surveillance for Any Reason
Description: Percentage of patients exiting active surveillance for any reason will be computed along with its 95% confidence interval.
Time Frame: At 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Apalutamide
Number analyzed (Participants) | 22
Percentage of participants | 22.7 [9.3 to 45.9]

4. Secondary Outcome: Percent of Men Undergoing Local Treatment
Description: Computed along with its 95% confidence interval.
Time Frame: At 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Apalutamide
Number analyzed (Participants) | 19
Participants | 5

5. Secondary Outcome: Local Treatment Free Survival
Description: Median treatment free survival will be estimated using Kaplan-Meier methods and 95% confidence interval will be calculated
Time Frame: Up to 730 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apalutamide
Number analyzed (Participants) | 22
days | 874 [805 to 9999]

6. Secondary Outcome: Prostate-specific Antigen Progression Rate
Description: Prostate-specific antigen progression rate is the proportion of patients that had PSA progression following treatment. PSA progression is as a confirmed rising prostate-specific antigen >= 2 ng/mL, with subsequent PSA values obtained at least one week apart.
Time Frame: At 2 years
Measure: Number; unit: Percentage of participants
Arm/Group | Apalutamide
Number analyzed (Participants) | 22
Percentage of participants | 100

7. Secondary Outcome: Prostate-specific Antigen Progression Free Survival as Defined by the Prostate Cancer Working Group 2 Criteria
Description: Prostate-specific antigen progression free survival will be estimated using Kaplan-Meier methods and 95% confidence interval will be estimated using Greenwood's formula.
Time Frame: At 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apalutamide
Number analyzed (Participants) | 22
days | 365 [204 to 401]

8. Secondary Outcome: Change in Radiographic Disappearance of Magnetic Resonance Imaging Detectable Prostate Cancer
Description: This calculates the percentage of participants with radiographic disappearance of magnetic resonance imaging detectable prostate cancer. This is only in patients with a baseline nodule that is Prostate Imaging Reporting and Data System 3 or more and > 5 mm.
Time Frame: Baseline to up to 90 days
Population: Only 1 patient had paired MRI at baseline and again at post-treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Apalutamide
Number analyzed (Participants) | 1
percentage of participants | 0

9. Secondary Outcome: Change in Quality of Life: FACT-P Assessment
Description: As assessed using the Functional Assessment of Cancer Therapy-Prostate (FACT-P) surveys. Functional Assessment of Cancer Therapy-Prostate is a validated quality of life survey specific for patients with prostate cancer. The total FACT-P score ranges from 0 to 156, with higher scores indicating better quality of life. The change in FACT-P score between baseline and day 730 is reported.
Time Frame: Baseline compared to 730 days
Population: Only 14 subjects completed Day 730 survey.
Measure: Median (Inter-Quartile Range); unit: Change in median FACT-P score
Arm/Group | Apalutamide
Number analyzed (Participants) | 14
Change in median FACT-P score | 3.17 [-3 to 9]

10. Secondary Outcome: Change in Quality of Life: SF-36 Physical Functioning
Description: As assessed using the Short Form-36 (SF-36) survey physical functioning subscale. Short Form-36 is a validated quality of life survey. This is a generic survey to assess an individual's overall well-being, and is not specific to one disease. The SF-36 physical functioning subscale score ranges from 0 to 100, with higher scores indicating better quality of life. The change in SF-36 energy/fatigue subscale score between baseline and day 730 is reported.
Time Frame: Baseline compared to 730 days
Population: Only 14 subjects completed Day 730 survey.
Measure: Median (Inter-Quartile Range); unit: Change in median SF-36 subscale score
Arm/Group | Apalutamide
Number analyzed (Participants) | 14
Change in median SF-36 subscale score | -17.65 [.50 to 50]

11. Secondary Outcome: Change in Quality of Life: SF-36 Energy/Fatigue
Description: As assessed using the Short Form-36 (SF-36) survey energy/fatigue subscale. Short Form-36 is a validated quality of life survey. This is a generic survey to assess an individual's overall well-being, and is not specific to one disease. The SF-36 energy/fatigue subscale score ranges from 0 to 100, with higher scores indicating better quality of life. The change in SF-36 energy/fatigue subscale score between baseline and day 730 is reported.
Time Frame: Baseline compared to 730 days
Population: Only 14 subjects completed Day 730 survey.
Measure: Median (Inter-Quartile Range); unit: Change in median SF-36 subscale score
Arm/Group | Apalutamide
Number analyzed (Participants) | 14
Change in median SF-36 subscale score | 12.5 [-5 to 20]

12. Secondary Outcome: Change in Quality of Life: SF-36 Emotional Well Being
Description: As assessed using the Short Form-36 (SF-36) survey emotional well being subscale. Short Form-36 is a validated quality of life survey. This is a generic survey to assess an individual's overall well-being, and is not specific to one disease. The SF-36 emotional well being subscale score ranges from 0 to 100, with higher scores indicating better quality of life. The change in SF-36 emotional well being subscale score between baseline and day 730 is reported.
Time Frame: Baseline compared to 730 days
Population: Only 14 subjects completed Day 730 survey.
Measure: Median (Inter-Quartile Range); unit: Change in median SF-36 subscale score
Arm/Group | Apalutamide
Number analyzed (Participants) | 14
Change in median SF-36 subscale score | 6 [-4 to 24]

ADVERSE EVENTS:
Time Frame: Through study completion, which corresponded to a median time of 753 days.
Arm/Group | Apalutamide
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 23/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apalutamide (N=23)
Nausea (Gastrointestinal disorders) | 2 (2)
Hot Flashes (Vascular disorders) | 5 (5)
Hypothyroidism (Endocrine disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 7 (7)
Fatigue/Decreased Energy (General disorders) | 18 (18)
Insomnia (Psychiatric disorders) | 2 (2)
Libido Decreased (Psychiatric disorders) | 5 (5)
Labile Mood (Psychiatric disorders) | 1 (1)
Cognitive Disturbance (Psychiatric disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Nipple Sensitivity/Tenderness (Reproductive system and breast disorders) | 11 (11)
Flu Like Symptoms (General disorders) | 1 (1)
Weight Loss/Anorexia (Metabolism and nutrition disorders) | 5 (7)
Mastodynia (Reproductive system and breast disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3)
Rhinorrhea (Infections and infestations) | 1 (1)
Increased/Elevated TSH (Investigations) | 4 (4)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Memory Impairment/Forgetfulness/Amnesia (Psychiatric disorders) | 3 (3)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Shingles (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Edema (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Bowel Movement Frequency (Gastrointestinal disorders) | 1 (1)
Lower Urinary Tract Symptoms (Renal and urinary disorders) | 2 (2)
Sinusitis (Immune system disorders) | 1 (1)
Tingling (Nervous system disorders) | 1 (1)
Brain Fog (Psychiatric disorders) | 1 (1)
Postural Dizziness/Balance Changes (Nervous system disorders) | 4 (4)
Concentration Impairment (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3)
Muscositis Oral (Gastrointestinal disorders) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dribbling (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Breast Tenderness (Reproductive system and breast disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 2 (2)
Lack of Body Odor (Skin and subcutaneous tissue disorders) | 1 (1)
Ejaculation Disorder (Reproductive system and breast disorders) | 1 (1)
Burning Sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Decreased Mental Acuity (Psychiatric disorders) | 1 (1)
Cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Nipple Itchiness (Reproductive system and breast disorders) | 1 (1)
Warmer Body (Vascular disorders) | 2 (2)
Akathisia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1)
Sore Throat (Immune system disorders) | 1 (1)
Painful Callus Bumps (Skin and subcutaneous tissue disorders) | 1 (1)
Upper Respiratory Infection Symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Impaired Vision (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Perceived Shrinking of Genitals (Reproductive system and breast disorders) | 1 (1)
Testicle Pain (Reproductive system and breast disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Bronchitis (Reproductive system and breast disorders) | 1 (1)
Chest Tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Clostridium Difficile Enteritis (Gastrointestinal disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
We acknowledge that the small sample size of this study is one of its primary limitations, which was further challenged by its premature termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT02721979/Prot_SAP_001.pdf
  • Informed Consent Form (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT02721979/ICF_000.pdf